CLINICAL TRIAL: NCT02821351
Title: Advanced Cardiac Therapeutics DiamondTemp TempeRAture-Controlled and Contact Sensing RF Ablation Clinical Trial for Atrial Fibrillation
Brief Title: ACT DiamondTemp TempeRAture-Controlled and Contact Sensing RF Ablation Clinical Trial for Atrial Fibrillation
Acronym: TRAC-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTAF-CZ01
Record Dates: First submitted 2016-06-22; First posted 2016-07-01 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Afib
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DiamondTemp (Experimental): Bilateral pulmonary vein isolation by RF ablation using DiamondTemp temperature controlled catheter and RF generator/pump system
  Interventions: Device: Radio frequency (RF) Cardiac ablation

INTERVENTIONS:
Device: Radio frequency (RF) Cardiac ablation — Catheter based RF cardiac ablation to treat Paroxysmal Atrial Fibrillation
  Other Names: RF Ablation

SUMMARY:
The primary objective of this study is to establish the safety and performance effectiveness of the DiamondTemp System for the treatment of drug refractory, recurrent, symptomatic paroxysmal atrial fibrillation (PAF).

DETAILED DESCRIPTION:
Study Title: Advanced Cardiac Therapeutics DiamondTemp TempeRAture-Controlled and Contact Sensing RF Ablation Clinical Trial for Atrial Fibrillation: TRAC-AF

Sponsor: Advanced Cardiac Therapeutics 2880 Lakeside Drive Suite 250 Santa Clara, CA 95054

Protocol No: DTAF-CZ01

Product: Cardiac Ablation Catheter and RF Generator/Pump System Investigational Device: DiamondTemp System (Inclusive of the DiamondTemp Ablation Catheter, DiamondTemp Catheter-to-RFG Cable, DiamondTemp GenConnect Cable, DiamondTemp RF Generator, DiamondTemp Irrigation Pump and DiamondTemp Irrigation Tubing)

PROTOCOL SUMMARY Advanced Cardiac Therapeutics DiamondTemp TempeRAture-Controlled and Contact Sensing RF Ablation Clinical Trial for Atrial Fibrillation: TRAC-AF

Study Objective:

The primary objective of this study is to assess the safety and performance effectiveness of the DiamondTemp System for the treatment of drug refractory, recurrent, symptomatic paroxysmal atrial fibrillation (PAF).

Investigational Device:

The investigational device in this clinical study is the DiamondTemp System inclusive of

* DiamondTemp Catheter (UPN: CZDT100S, CZDT100L)
* DiamondTemp Catheter-to RFG Cable (UPN: CZDC100)
* DiamondTemp GenConnect Cable (UPN: CZDTGC100)
* DiamondTemp RF Generator (UPN:CZDTG100)
* DiamondTemp Irrigation Pump (UPN: CZDP100)
* DiamondTemp Irrigation Tubing Set (UPN: CZDTS100)

System Accessories:

* Dispersive Indifferent Patch (DIP) electrodes
* Power Cord
* EGM Cable (not supplied)
* St. Jude Maestro GenConnect (not supplied)

The investigational device can be used with commonly available EP Recording System, Cardiac Stimulator and the ST. Jude EnSite™ Velocity™ Cardiac Mapping System.

There are no control devices in this study.

Study Design/Planned Number of Subjects/Number of Centers This study is a prospective, single center, single arm study. A maximum of 75 subjects will be enrolled in the study to include a maximum of 5 roll-in subjects in one investigational center in the Czech Republic.

Primary Endpoints The primary endpoint events for this trial as follows are to assess the safety and performance effectiveness of the DiamondTemp System for the treatment of drug refractory, recurrent, symptomatic PAF.

* Primary Safety Endpoint: The safety of the DiamondTemp System will be assessed by evaluating the nature and frequency of serious adverse events (SAE) and serious adverse device effects (SADE) during the time of the ablation procedure and within 7 days afterwards.
* Primary Effectiveness Endpoint: The effectiveness of the DiamondTemp System will be evaluated post-ablation with demonstration of acute procedural success defined as isolation of clinically relevant pulmonary veins by demonstration of block or isolation of signals confirmed after delivery of the ablation treatment. Depending on EP lab protocol, one method will be chosen.

Secondary Endpoints

The following secondary endpoint will be evaluated to support the results of the primary endpoints:

• Secondary Safety Endpoint: The chronic safety of the DiamondTemp System will be assessed by evaluating the nature and frequency of adverse events (AE) and adverse device effects (ADE) at 30 days, 90 days, 6 months and 12 months post-procedure.

Study Duration The duration of the study is expected to last approximately 18 months from the first enrollment to final report for assessment of endpoints. An additional 12 months to the study closeout after the last follow-up.

Key Inclusion Criteria

* Suitable candidate for intra-cardiac mapping for arrhythmias
* History of recurrent symptomatic PAF WITH ≥2 episodes reported within the 365 days (12) months prior to enrollment
* At least 1 episode of atrial fibrillation (AF) documented by Holter monitor, rhythm strip, trans-telephonic monitor (TTM), or 12-lead ECG prior to enrollment
* Refractory to at least one Class I-IV anti-arrhythmic drug (AAD)
* Eighteen (18) years of age or above
* Competent and willing to provide written informed consent to participate in the study and agree to comply with the follow-up visits and evaluation

Key Exclusion Criteria

* Previous ablation procedure in the left atrium
* Intracardiac thrombus, tumor or other abnormality that precludes catheter introduction and placement
* Known severe cerebrovascular disease or history of cerebrovascular event (within 1 month)
* Cardiac surgery within the past two months.
* Short life expectancy (< 1 yr.) due to other illnesses, such as cancer or pulmonary, hepatic, or renal disease
* Uncontrolled congestive heart failure (NYHA Class III or IV)
* Unstable angina or acute myocardial infarction within the past three months
* Bleeding, clotting disorders, or known thrombosis
* Heart valve replacement
* Mitral clip (Evalve)
* Unable or unwilling to take anti-coagulants

Ablation Procedure The ablation procedure will consist of documentation of pre-ablation pulmonary vein (PV) potentials, conducting PV isolation using the DiamondTemp System, providing documentation of PV entrance block. Investigator can opt to perform other ablations if any non- PV foci are involved in atrial arrhythmia.

Follow-up Schedule

* Screening visit any time during six (6) months before ablation procedure
* Ablation Procedure (Day 0, all follow-ups post ablation are based on this date)
* Discharge (5-72 hours)
* 7-Day Phone Check (7 + 3 days)
* 1-Month Follow-up (30 + 5 days)
* Repeat Mapping Procedure
* Repeat Ablation Procedure, if necessary
* 3-Month Follow-up (90 + 10 days)
* 6-Month Follow-up (180 + 30 days)
* 12-Month Follow-up (365 + 30 days)
* Additional Follow-up visits (as determined necessary)

The study will be considered complete for the purpose of reporting results with regards to the primary endpoints after all subjects have completed the 7-Day follow-up. A final study closeout report will be created after the last 12-month follow-up visit.

ELIGIBILITY:
Study Inclusion Criteria

Subjects for this study must meet ALL of the following criteria:

* Suitable candidate for intra-cardiac mapping and ablation for arrhythmias.
* History of recurrent symptomatic PAF1 WITH ≥2 episodes reported within the 365 days (12) months prior to enrollment.
* At least one episode of AF documented by Holter monitor, rhythm strip, trans-telephonic monitor (TTM), or 12-lead ECG prior to enrollment
* Refractory to at least one Class I - IV anti-arrhythmic drug (AAD)
* Eighteen (18) years of age or above
* Competent and willing to provide written informed consent to participate in the study and agree to comply with the follow-up visits and evaluation.

Study Exclusion Criteria

Candidates will be excluded from the study if any of the following conditions apply:

* Previous left atrial ablation procedure
* Intracardiac thrombus, tumor or other abnormality that precludes catheter introduction and placement
* Known severe cerebrovascular disease or history of cerebrovascular event (within 1 month)
* Patients with severely impaired kidney function as measured by a Cockcroft-Gault Glomerular Filtration Rate (GFR)3 with a GFR ≤ 29. This is calculated as follows for males:

GFR = (140 - age) x weight x .85 (for females) PCr x 72 where age is specified in years, weight in kg, and PCr is Serum Creatinine in mg/dL Female GFR is reduced by 15% of the above calculated value for males.

* Active gastrointestinal bleeding
* Active infection or fever (> 100.5 F/38 C)
* Sepsis
* Cardiac surgery within the past two months
* Short life expectancy (< 1yr) due to other illnesses, such as cancer or pulmonary, hepatic, or renal disease
* Significant anemia (hemoglobin < 8.0 mg/dL)
* Severe uncontrolled systemic hypertension (systolic press. > 240 mm Hg within the last 30 days)
* Documented anaphylaxis during previous exposure to angiographic contrast media
* Uncontrolled congestive heart failure (NYHA Class III or IV)
* Unstable angina or acute myocardial infarction within the past three months
* Bleeding, clotting disorders, or known thrombosis
* Severe Peripheral vascular disease
* Uncontrolled diabetes
* Rheumatic heart disease
* Heart valve replacement
* Mitral clip (Evalve)
* Women who are of childbearing potential who are currently pregnant or not willing to use contraception for the duration of the study
* Active participation in another investigational protocol currently or the last 30 days
* Unable or unwilling to take anti-coagulants
* Unwilling or unable to comply with any protocol or follow up requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Nature and frequency of serious adverse events (SAE) and serious adverse device effects (SADE) | Seven days
  The safety of the DiamondTemp System will be assessed by evaluating the nature and frequency of serious adverse events (SAE) and serious adverse device effects (SADE) during the time of the ablation procedure and within 7 days afterwards.
Electrical Isolation of treated Pulmonary Vein from Left Atrium | Seven days
  The effectiveness of the DiamondTemp System will be evaluated post-ablation with demonstration of acute procedural success defined as isolation of clinically relevant pulmonary veins by demonstration of block or isolation of signals confirmed after delivery of the ablation treatment. Depending on EP lab protocol, one method will be chosen.

SECONDARY OUTCOMES:
Nature and frequency of serious adverse events (SAE) and serious adverse device effects (SADE) up to a year after treatment | During 12 months after the treatment
  The chronic safety of the DiamondTemp System will be assessed by evaluating the nature and frequency of adverse events (AE) and adverse device effects (ADE) at 30 days, 90 days, 6 months and 12 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, MD, PhD, Principal Investigator — Na Homolce Hospital
Locations (4):
- Czechia (3):
  - St Anne's University Hospital, Brno
  - Institut Klinické a Experimentální Medicíny (IKEM), Prague
  - Nemocnice Na Homolce, Prague
- Clinique Pasteur, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Starek Z, Lehar F, Jez J, Pesl M, Neuzil P, Sediva L, Petru J, Dujka L, Funasako M, Kautzner J, Peichl P, Aldhoon B, Albenque JP, Combes S, Boveda S, Dukkipati SR, Reddy VY. Efficacy and safety of novel temperature-controlled radiofrequency ablation system during pulmonary vein isolation in patients with paroxysmal atrial fibrillation: TRAC-AF study. J Interv Card Electrophysiol. 2022 Aug;64(2):375-381. doi: 10.1007/s10840-021-00986-0. Epub 2021 Jun 5. PMID 34089431
- [Derived] Iwasawa J, Koruth JS, Petru J, Dujka L, Kralovec S, Mzourkova K, Dukkipati SR, Neuzil P, Reddy VY. Temperature-Controlled Radiofrequency Ablation for Pulmonary Vein Isolation in Patients With Atrial Fibrillation. J Am Coll Cardiol. 2017 Aug 1;70(5):542-553. doi: 10.1016/j.jacc.2017.06.008. PMID 28750697